CLINICAL TRIAL: NCT04623645
Title: Ultrasound Guided Bilateral Superior Laryngeal Nerve Block Compared With Blind Block Technique For Awake Fibre-optic Intubation In Suspected Difficult Intubation
Brief Title: Ultrasound Guided Superior Laryngeal Nerve Block Compared With Blind Block Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Alshaymaa Mortada Ali Eltohry, clinical researcher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MS 19/ 2020
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Airway Complication of Anesthesia
Keywords: Suspected Difficult Intubation
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound group (Experimental): patient using ultrasound technique.probe will be placed over submandibular area, the thyrohoid muscle and thyrohyoid membrane will be identified between greater horn fo hyoid bone and thyroid cartilage , 3 ml of lignocaine will be placed on space between thim and the procedure will repeated on contra lateral side.
  Interventions: Device: ultrasound technique
- anatomical blind group (Active Comparator): patient using anatomical land mark technique, internal branch of superior laryngeal nerve will be blocked slightly anterior to greater horn of hyoid bone . by 3 ml lignocaine . the procdure will be repeated on contra lateral side .
  Interventions: Device: ultrasound technique

INTERVENTIONS:
Device: ultrasound technique — evaluate the effect of ultrasound guided technique for block of internal branch of superior laryngeal nerve

SUMMARY:
The aim of this study is to evaluate the effect of ultrasound guided technique for block of internal branch of superior laryngeal nerve in surgical patient in comparison to blind anatomical technique.

DETAILED DESCRIPTION:
Airway anesthesia is pivotal for successful awake intubation provided either topically or by nerves blocks. Airway blocks are technically harder to perform with more complications possibilities. However, in experienced hands, they can be useful as they provide better intubating conditions.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists ( ASA ) physical status I and II.
2. Age between 40-60 years.
3. Modified Mallampati class III-IV .

Exclusion Criteria:

1. Local pathology of the neck.
2. Bleeding diathesis.
3. Allergy to local anesthetic agent.
4. Intellectual impairment.
5. Psychiatric disease.
6. Body mass index ≥30 kg/m2.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
assessment the quality of airway anesthesia | Up to 2 years post baseline
  The Quality of Airway anesthesia will be graded as: 0 = no coughing or gagging in response to intubation, 1 = mild coughing or gagging that will not hinder intubation, 2 = moderate coughing or gagging that will interfere minimally with intubation,3 = severe coughing or gagging that make intubation difficult and 4 = very severe coughing or gagging that will require additional local anesthetic or change in technique to achieve successful intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Mohamed Shafik, professor, Study Chair — Ain shams university, faculty of medicine; Abeer Mohamed Abdel-Aziz, professor, Study Director — Ain shams university, faculty of medicine
Locations (1):
- Alshaymaa Mortada Ali Eltohry, Alexandria, Please Select An Option, Egypt

REFERENCES:
- [Background] Manikandan S, Neema PK, Rathod RC. Ultrasound-guided bilateral superior laryngeal nerve block to aid awake endotracheal intubation in a patient with cervical spine disease for emergency surgery. Anaesth Intensive Care. 2010 Sep;38(5):946-8. doi: 10.1177/0310057X1003800523. PMID 20865885
- [Background] Ramkumar V. Preparation of the patient and the airway for awake intubation. Indian J Anaesth. 2011 Sep;55(5):442-7. doi: 10.4103/0019-5049.89863. PMID 22174458